CLINICAL TRIAL: NCT01620112
Title: The Effects of Different Clonidine Concentrations on Axillary Brachial Plexus Block With 1,5% Lidocaine for Upper Limb Surgery: a Prospective Randomized Study
Brief Title: The Effects of Different Clonidine Concentrations on Axillary Brachial Plexus Block With 1,5% Lidocaine
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Universidade Federal do Rio de Janeiro (Other)
Responsible Party: Principal Investigator, Alexandra Rezende Assad, Assad AR, Universidade Federal do Rio de Janeiro
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 090/2002
Record Dates: First submitted 2012-06-09; First posted 2012-06-15 (Estimated); Last update posted 2012-06-15 (Estimated); Status verified 2012-06

CONDITIONS: Fascicular Block; Motor Activity; Pain, Postoperative; Latency Period
Keywords: brachial plexus; lidocaine; alfa 2 adrenergic receptor clonidine; orthopedic procedure
MeSH Terms: conditions — Bundle-Branch Block; Motor Activity; Pain, Postoperative | interventions — Lidocaine

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- low clonidine concentration (Active Comparator): clonidine concentration 1 ml on 40 ml of lidocaine 1.5% for upper brachial plexus
  Interventions: Drug: low clonidine concentration
- lidocaine 20 ml 1,5% (Active Comparator): lidocaine 20 ml 1,5% without clonidine for axillary brachial plexus block for upper limb surgery
  Interventions: Drug: Lidocaine
- high clonidine concentration (Active Comparator): clonidine concentration 150 mcg on 20 ml of lidocaine 1,5% for upper brachial plexus
  Interventions: Drug: high Clonidine concentration
- 40 ml lidocaine 1,5% (Active Comparator): 40 ml of lidocaine 1,5% without clonidine for upper brachial plexus
  Interventions: Drug: Lidocaine 40 ml

INTERVENTIONS:
Drug: high Clonidine concentration — Clonidine 1 ml - 150 mcg on 20 ml de lidocaine 1,5% on axillary brachial plexus block for upper limb surgery
  Arms: high clonidine concentration
Drug: low clonidine concentration — Clonidine 1 ml - 150 mcg on 40 ml of lidocaine 1,5% - single injection on axillary brachial plexus block for upper limb
  Arms: low clonidine concentration
Drug: Lidocaine — Lidocaine 1,5% 20 ml 300 mg for single injection on axillary brachial plexus block for upper lim surgery
  Arms: lidocaine 20 ml 1,5%
Drug: Lidocaine 40 ml — Lidocaine 40 ml 1,5% 600 mg single injection for axillary brachial plexus block for upper limb surgery
  Arms: 40 ml lidocaine 1,5%

SUMMARY:
The purpose of this study is to determine whether different clonidine concentration on axillary brachial plexus block with 1,5% lidocaine for upper limb surgery may influence the sensory and motor block onset time and duration, postoperative analgesia duration, postoperative pain intensity

DETAILED DESCRIPTION:
Brachial plexus blocks are frequently used in surgical procedures involving the upper limb because they facilitate surgical anaesthesia, muscle relaxation and post-operative analgesics.

Various drugs are used to supplement local anaesthetics during brachial plexus block. Many studies in the literature show that clonidine, which is an alpha-2 agonist, prolongs the length of anesthesia and post-operative analgesia.4,5 However, clonidine's side effects-such as hypotension, bradycardia and sedation can limit its use.

There are no studies comparing different clonidine concentrations on the axillary brachial block, so the hypothesis of the present study was that different clonidine concentrations and LA volumes may influence the anaesthesia and analgesia quality on this type of regional block.

ELIGIBILITY:
Inclusion Criteria:

* both genders,
* over 18 years old,
* American Society of Anesthesiologists (ASA) 1 to 3

Exclusion Criteria:

* patients with chronic use of analgesics and non-steroidal anti-inflammatories drugs,
* pregnant,
* with infection at the puncture site,
* coagulopathies or intolerance to drugs used in the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2009-02; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
sensorial and motor block duration | 24 hours after surgery
  to compare two concentrations of clonidine on different volumes of lidocaine, in terms of sensorial and motor block duration

SECONDARY OUTCOMES:
adverse effects of additive clonidine on axillary brachial plexus block in upper limb surgery | 24 hours after surgery
  analyse the adverse effects of additive clonidine on axillary brachial plexus block in upper limb surgery
postoperative analgesia duration | 24 hours
  to compare two concentrations of clonidine on different volumes of lidocaine, in terms of postoperative analgesia duration
sensorial and motor block onset time | 24 hours
  to compare two concentrations of clonidine on different volumes of lidocaine, in terms of sensorial and motor block onset time
postoperative pain intensity | 24 hours
  to compare two concentrations of clonidine on different volumes of lidocaine, in terms postoperative pain intensity